CLINICAL TRIAL: NCT06882226
Title: Evaluation of the Emotional Burden of the Nurse in Onco-hematology
Brief Title: Evaluation of the Emotional Burden of the Nurse
Acronym: EMOCARE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7360
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maslach burnout inventory — Assessing the emotional burden on nursing staff

SUMMARY:
Asses the emotional burden on nursing staff and how much they are at risk for burnout.

DETAILED DESCRIPTION:
The study involves the administration of a questionnaire paper questionnaire (maslach burnout scale) in the presence.

ELIGIBILITY:
Inclusion Criteria:

* Nursing personnel afferent to the OU of hematology and stem cell transplantation hematopoietic and the uoc geriatric hematology and rare hemapathies with more than 2 years of experience in the above departments.
* Signature of informed consent.
* Ability to understand and complete.

Exclusion Criteria:

* Nursing staff not belonging to the departments of hematology
* Failure to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurse attached to uoc 1E hematology and TCSE and uoc 5E geriatric hematology and rare diseases.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of emotional burden on nursing staff | 1 month
  Maslach burnout scale

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Lamberti, Principal Investigator — FPG